CLINICAL TRIAL: NCT01452685
Title: A Phase II, Multicenter, Long-term Extension Study to Compare the Safety and Efficacy of TAK-385 (10, 20, and 40 mg) Following Oral Administration for 12 Weeks or More in the Treatment of Endometriosis
Brief Title: A Long-term Extension Study of TAK-385 in the Treatment of Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-385/OCT-101; U1111-1123-6973 (Registry Identifier: WHO); JapicCTI-11589 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-08-31; First posted 2011-10-17 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Endometriosis
Keywords: Drug Therapy
MeSH Terms: conditions — Endometriosis | interventions — relugolix; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- TAK-385 10 mg QD (Experimental)
  Interventions: Drug: TAK-385
- TAK-385 20 mg QD (Experimental)
  Interventions: Drug: TAK-385
- TAK-385 40 mg QD (Experimental)
  Interventions: Drug: TAK-385
- Leuplin (Other)
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: Placebo — TAK-385 placebo-matching tablets, orally, once daily and leuprorelin acetate placebo injection, subcutaneously, once every 4 weeks for up to 12 weeks.
  Arms: Placebo
Drug: TAK-385 — TAK-385 10 mg, tablets, orally, once daily and leuprorelin acetate placebo injection, subcutaneously, once every 4 weeks for up to 12 weeks.
  Arms: TAK-385 10 mg QD
Drug: TAK-385 — TAK-385 20 mg, tablets orally, once daily and leuprorelin acetate placebo injection, subcutaneously, once every 4 weeks for up to 12 weeks.
  Arms: TAK-385 20 mg QD
Drug: TAK-385 — TAK-385 40 mg, tablets, orally, once daily and leuprorelin acetate placebo injection, subcutaneously, once every 4 weeks for up to 12 weeks.
  Arms: TAK-385 40 mg QD
Drug: Leuprorelin acetate — TAK-385 placebo-matching tablets, orally, once daily and leuprorelin acetate 3.75 mg injection, subcutaneously, once every 4 weeks for up to 12 weeks
  Other Names: Leuplin
  Arms: Leuplin

SUMMARY:
The purpose of this study is to compare the long term safety and efficacy of TAK-385, once daily (QD) following continued administration in participants who completed a Phase II dose-finding study.

DETAILED DESCRIPTION:
This study is a long-term extension study for evaluation of the safety and efficacy of TAK-385 following administration for 24 weeks (calculated from Visit 3 in the TAK-385/CCT-101 study) in participants from the Phase II dose-finding study (TAK-385/CCT-101 study).

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have completed TAK-385/CCT-101 study

Exclusion Criteria:

1. Participants who had an adverse event in TAK-385/CCT-101 study which makes continued administration of the study drug difficult
2. Participants who became unable to comply with the protocol due to onset of a new disease, symptom, finding, or aggravation of clinical laboratory findings
3. Participants in whom investigator deems that the study drug shows no efficacy based on the level of pain, menstruation status, and the status of analgesic drug intake in TAK-385/CCT-101 study, or that study continuation represents an unacceptable risk
4. Participants in whom investigator deems that study continuation is difficult due to the occurrence of low estrogen symptoms in TAK-385/CCT-101 study which were attributed to the pharmacological effects of the study drug taking into account the level and frequency of the adverse events etc. as well as the risk-benefit of participants.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | Up to Week 24.
  Measured by Dual-energy X-ray absorptiometry (DXA)
Treatment-emergent Adverse Events | Up to Week 16
  Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through the last visit (Week 16)
Vital Signs | Up to Week 24
  Vital signs will include body temperature, sitting blood pressure and pulse (bpm).
Body Weight | Up to Week 24
Electrocardiograms | Up to Week 24.
Laboratory Values | Up to Week 24
Serum NTx | Up to Week 24
  NTx is one of the biochemical bone metabolism markers
Serum BAP | Up to Week 24
  BAP is one of the biochemical bone metabolism markers

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Score for Pelvic Pain | Up to Week 24
  Pelvic pain will be assessed using the VAS as pain evaluation scale
VAS Score for Dyspareunia | Up to Week 24
  Dyspareunia will be assessed using the VAS as pain evaluation scale

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (69):
- Japan (69):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Funabashi-shi, Chiba
  - Ichihara-shi, Chiba
  - Yachiyo-shi, Chiba
  - Nihama-shi, Ehime
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Iizuka-shi, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Yanagawa-shi, Fukuoka
  - Koriyama-shi, Fukushima
  - Takayama-shi, Gifu
  - Takasaki-shi, Gunma
  - Hirosima-shi, Hiroshima
  - Ebetsu-shi, Hokkaido
  - Ishikari-shi, Hokkaido
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Kako-gun, Hyōgo
  - Kawanishi-shi, Hyōgo
  - Kobe, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Marugame-shi, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Hiratsuka-shi, Kanagawa
  - Kamakura-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Yamato-shi, Kanagawa
  - Yokohama, Kanagawa
  - Nankoku-shi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Matsumoto-shi, Nagano
  - Nagano, Nagano
  - Suzaka-shi, Nagano
  - Nara, Nara
  - Ōita, Oita Prefecture
  - Kurashiki-shi, Okayama-ken
  - Okayama, Okayama-ken
  - Hirakata-shi, Osaka
  - Ibaraki-shi, Osaka
  - Ikeda-shi, Osaka
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Suita-shi, Osaka
  - Tondabayashi-shi, Osaka
  - Toyonaka-shi, Osaka
  - Iruma-shi, Saitama
  - Kusatsu-shi, Shiga
  - Hamamatsu, Shizuoka
  - Numazu-shi, Shizuoka
  - Yaizu-shi, Shizuoka
  - Komatsushima-shi, Tokushima
  - Naruto-shi, Tokushima
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Machida-shi, Tokyo
  - Minato-ku, Tokyo
  - Ohta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Suginami-ku, Tokyo
  - Toyama, Toyama
  - Yamaguchi, Yamaguchi

REFERENCES:
- [Derived] Osuga Y, Seki Y, Tanimoto M, Kusumoto T, Kudou K, Terakawa N. Relugolix, an oral gonadotropin-releasing hormone (GnRH) receptor antagonist, in women with endometriosis-associated pain: phase 2 safety and efficacy 24-week results. BMC Womens Health. 2021 Jun 21;21(1):250. doi: 10.1186/s12905-021-01393-3. PMID 34154590